CLINICAL TRIAL: NCT01952236
Title: Web and Mobile Smoking Cessation Interventions
Brief Title: Web and Mobile Smoking Cessation
Acronym: MobileQuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA172205-01
Record Dates: First submitted 2013-07-25; First posted 2013-09-27 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Smoking
Keywords: Smoking; Quit; Tobacco; Abstinence; Adult; Text Messaging; Web-based; Mobile phone; smartphone; internet; web
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web+Mobile (Experimental): A best-practices Web-based smoking cessation program integrated with a tailored treatment program delivered using a smartphone application.
  Interventions: Behavioral: Web+Mobile
- Web Only (Active Comparator): A best-practices Web-based smoking cessation program.
  Interventions: Behavioral: Web Only

INTERVENTIONS:
Behavioral: Web+Mobile — We propose to evaluate the efficacy and acceptability of a Web+Mobile tobacco cessation intervention in a 2-arm Randomized Controlled Trial with 1,271 adult study participants who agree to quit smoking within a pre-specified amount of time. Participants who meet eligibility criteria will be randomly assigned to either (a) an enhanced Web Only intervention or (b) an enhanced Web+Mobile intervention.
  Arms: Web+Mobile
Behavioral: Web Only — A Web-based PC-delivered best practices smoking cessation intervention.
  Arms: Web Only

SUMMARY:
This study seeks to develop and then perform a controlled efficacy Randomized Controlled Trial assessing tobacco abstinence of a best-practices Web-based PC-delivered smoking cessation intervention (QuitOnline) compared to a Mobile Smartphone-delivered intervention (MobileQuit). Study participants are randomized to one of two conditions: a Web Only intervention and the Web+Mobile intervention. The hypothesis is that the Web+Mobile approach will yield greater efficacy than the Web Only condition.

DETAILED DESCRIPTION:
The primary aims of this project are to:

1. Use an iterative formative development process to create two separate Web-based smoking cessation programs (Web+Mobile, Web Only).
2. Compare the efficacy of the two smoking cessation programs in terms of tobacco abstinence. The investigators hypothesize that the Web+Mobile condition will be significantly more efficacious in terms of tobacco abstinence than the Web Only condition.
3. Evaluate program usage/participant engagement, treatment acceptability, and consumer satisfaction. The investigators hypothesize that both conditions will be acceptable and that the Web+Mobile condition will have significantly greater usage and higher consumer satisfaction than the Web Only condition.

The secondary aims of this proposal are to:

1. Evaluate the differences between conditions on ancillary tobacco outcomes. The investigators hypothesize that the participants assigned to the Web+Mobile condition who continue to smoke will nonetheless report a greater decline in the smoking rate and more quit attempts.
2. Evaluate predictors and condition moderators of tobacco abstinence. The investigators will conduct exploratory analyses of the association of treatment outcomes to participant characteristics (e.g., baseline smoking rate, nicotine dependence level, partner's tobacco use, prior quitting attempts, prior use of pharmacological adjuncts, and other demographic factors).
3. Evaluate putative mechanisms of change. The investigators will test whether change in the putative mechanisms of change (i.e., self-efficacy, program use, use of pharmacological adjuncts) mediate the association between the intervention condition and 3-month sustained abstinence from the 3 month to 6 month assessments.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Cigarettes are primary tobacco of use
* Smoke ≥ 5 cigs/day for the previous 6 months
* Want to quit in next 14 days
* Use a smartphone and willing to potentially receive/send up to 150 text messages over the six months of the program
* Access to the Internet
* Have a valid personal e-mail address
* Be a U.S. citizen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1266 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in all-tobacco abstinence from enrollment to 3 months and 6 months post enrollment | Change from enrollment to 3 months and 6 months post enrollment
  Change in all-tobacco abstinence from enrollment to 3 and 6 months. Measured using 7 day point prevalence.

SECONDARY OUTCOMES:
Program usage, treatment acceptability, consumer satisfaction 3 months post enrollment follow-up | 3 months post enrollment
  Evaluate program usage of each condition using unobtrusive measures of website visits (both conditions: number, duration, webpages viewed, interactive activities used), use of mobile intervention components (Web+Mobile condition only: number of calls received, number of responses received, extent of data collected), treatment acceptability, and consumer satisfaction
Predictors and condition moderators of tobacco abstinence at 6-months follow-up | Baseline to 6-month follow-up
  Analyses of the association of primary outcomes to participant characteristics (e.g., baseline smoking rate, nicotine dependence level, partner's tobacco use, prior quitting attempts, prior use of pharmacological adjuncts, and other demographic factors).

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Danaher, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Danaher BG, Tyler MS, Crowley RC, Brendryen H, Seeley JR. Outcomes and Device Usage for Fully Automated Internet Interventions Designed for a Smartphone or Personal Computer: The MobileQuit Smoking Cessation Randomized Controlled Trial. J Med Internet Res. 2019 Jun 6;21(6):e13290. doi: 10.2196/13290. PMID 31172967
- See also: Oregon Research Institute — http://www.ori.org